CLINICAL TRIAL: NCT04174105
Title: A Phase 1/2, Open-Label, Ascending-Dose Clinical Study to Evaluate the Safety and Preliminary Efficacy of AT845, an AAV8-Delivered Gene Transfer Therapy in Patients With Late Onset Pompe Disease
Brief Title: Gene Transfer Study in Patients With Late Onset Pompe Disease
Acronym: FORTIS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT845-01; 2019-003595-38 (EudraCT Number)
Record Dates: First submitted 2019-11-13; First posted 2019-11-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pompe Disease (Late-onset)
Keywords: LOPD
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Intervention Model Description: Up to 3 nominal dose levels of AT845 are planned to be evaluated in this study. A single AT845 administration via IV infusion is planned for each subject. The initial dosing cohort received a single dose of 3×10^13 vg/kg. The second dose cohort will receive a single dose of 6×10^13 vg/kg. The third dose cohort will receive a single dose of 1×10^14 vg/kg. Dose escalation between cohorts will be based on evaluations of safety and in consultation with the independent DMC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Initial Dose Cohort (Experimental): 3x10^13 vg/kg of AT845 administered via intravenous infusion
  Interventions: Genetic: zocaglusagene nuzaparvovec
- Second Dose Cohort (Experimental): 6x10^13 vg/kg of AT845 administered via intravenous infusion
  Interventions: Genetic: zocaglusagene nuzaparvovec
- Third Dose Cohort (Experimental): 1x10^14 vg/kg of AT845 administered via intravenous infusion
  Interventions: Genetic: zocaglusagene nuzaparvovec

INTERVENTIONS:
Genetic: zocaglusagene nuzaparvovec — AT845 is an AAV8 vector delivering a functional copy of the human GAA gene, under the control of a muscle-specific promoter
  Other Names: AT845

SUMMARY:
This is a phase 1/2 open-label, ascending dose, multicenter clinical study to evaluate the safety and efficacy of AT845 in adult (aged ≥ 18 years) subjects, ambulatory or nonambulatory, with Late Onset Pompe Disease (LOPD).

DETAILED DESCRIPTION:
This study (FORTIS) will evaluate the safety and efficacy of an investigational gene replacement therapy, AT845, in adult subjects with LOPD. Subjects will receive a single dose of AT845 delivered via intravenous (IV) infusion.

Up to 3 nominal dose levels of AT845 are planned to be evaluated in this study. A single AT845 administration via IV infusion is planned for each subject. The initial dosing cohort received a single dose of 3x10^13 vg/kg of AT845. The second dose cohort will receive a single dose of 6×10^13 vg/kg. The third dose cohort will receive a single dose of 1×10^14 vg/kg. Dose escalation between cohorts will be based on evaluations of safety and in consultation with the independent DMC.

There will be a core observation period of 48 weeks with scheduled visits and assessments. Following the conclusion of the core observation period, subjects will be seen every 6 months for a safety follow-up visit for up to 10 years postdose.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged ≥ 18 years.
* Participant has a documented clinical diagnosis of Pompe disease by genetic testing.
* Participant has received enzyme replacement therapy (ERT) with rhGAA for the previous ≥ 2 years.
* Participant has been on a stable standard dose (at least 20 mg/kg every 2 weeks) of ERT with rhGAA for at least the previous 6 months.
* Participant or legally authorized representative(s) (LAR) (if applicable) provides written informed consent.
* Participant and LAR(s) are willing and able to comply with study visits and study procedures.
* Participant must agree to refrain from blood or blood products donation and sperm or egg donation from the time of AT845 administration until the later of 90 days or 3 consecutive negative viral shedding samples
* Participants enrolled in previous protocol versions 1 through 9: Participant has upright FVC ≥ 30% of predicted normal value. Participants enrolled starting with protocol version 10 and subsequent amendments: Participant has upright FVC ≥ 30% and ≤ 85% of predicted normal value.
* Participants enrolled starting with protocol version 10 and subsequent amendments: Participant who is able to ambulate ≥ 40 m without stopping and without the use of an assistive device. The use of an assistive device for community ambulation is acceptable. (Participants enrolled under previous protocol versions 1 through 9 will not be excluded if they do not meet this criterion during Rescreening visit).

Exclusion Criteria:

* Participant is currently participating in an interventional study or has received gene or cell therapy.
* Participant tests positive for AAV8 antibodies with titers >1:20 neutralizing.
* Participant has received immune-modulating agents within 90 days before dosing (use of inhaled corticosteroids is allowed); use of other concomitant medications to manage chronic conditions must have been stable for at least 30 days before dosing. Concomitant medications that may predispose the participant to peripheral neuropathy will be evaluated.
* Participant has any clinically significant laboratory values (other than those directly associated with LOPD [e.g., GAA, serum creatine kinase (CK)]) that would preclude participation in the study.
* Participant has serological or viral load evidence of HIV-1 or HIV-2.
* Participant has received drugs for treatment of myopathy or neuropathy with immunosuppressive therapy (e.g., corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, IV immunoglobulin, rituximab) within 3 months prior to starting the study
* Participant has a high risk for a severe allergic reaction to rhGAA (ie, previous moderate to severe anaphylactic reaction to alglucosidase alfa or and/or a history of sustained high immunoglobulin G [IgG] antibody titers to alglucosidase alfa that suggests a high risk for an allergic reaction to ERT).
* Participant has a history of hypersensitivity to β2 agonist drugs such as albuterol, levalbuterol, bitolterol, pirbuterol, terbutaline, salmeterol, which contraindicates pulmonary function testing.
* Participant has an active viral infection based on clinical observation.
* Participant has a history of or concurrent medical condition other than Pompe disease that could jeopardize safety of the participant or impact study results.
* Participant has a history of, or currently has, a clinically important cardiac condition, such as an echocardiogram (ECHO) with ejection fraction below 40% or has symptoms or signs of cardiomyopathy that precludes enrollment.
* Participant has a contraindication to study drug or to corticosteroids, or has demonstrated hypersensitivity to any of the components of the study drug.
* Participant tests positive for GAA antibodies with titers > 1:50,000 total
* Participant has a history of hypersensitivity to MRI contrast agents including gadolinium.
* Participant has a known hypersensitivity to local anesthetics such as lidocaine.
* Participant has a bleeding diathesis, e.g., due to anti-coagulation or anti-platelet treatments.
* Participant has a concurrent medical condition (including uncontrolled diabetes, alcohol use disorder, certain autoimmune conditions, Lyme disease, active malignancy requiring chemotherapy and/or radiation, uremic nephropathy, known exposure to heavy metals) commonly associated with peripheral neuropathy. Other concurrent medical conditions that may predispose to peripheral neuropathy will be evaluated and action taken on a case-by-case basis, following discussion between the Investigator and Medical Monitor.
* Participant who is unwilling to withdraw from ERT.
* Participant has an active symptomatic large fiber peripheral neuropathy diagnosed by a neurologist at a screening visit.
* Age-related sensory changes on NCS without symptoms or mononeuropathy (refers to focal involvement of a single nerve, usually due to a local cause such as trauma, compression or entrapment) will not be excluded.
* Participant has clinically significant underlying liver disease at Screening, or has any of the following:
* Alanine Aminotransferase (ALT) > 2 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) > 2 × ULN
* Total bilirubin > 1.5 × ULN
* Alkaline phosphatase (ALP) > 2 × ULN
* ALT and AST are often higher than the normal range in Pompe disease patients. Participants whose liver laboratory tests fall outside the above ranges may be retested and, if the eligibility criteria are met on retesting, may be enrolled after confirmation by the Medical Monitor.
* In addition, participants with abnormal laboratory results related to confirmed benign liver conditions including Gilbert's syndrome (defined by asymptomatic unconjugated hyperbilirubinemia [17 to 70 µmol/L or 1 to 4 mg/dL]) and asymptomatic gallstones, will be considered eligible for the study notwithstanding their abnormal laboratory results and may be enrolled.
* Participant is currently on antiviral therapy for hepatitis B or C, or chronic/active hepatitis B or active hepatitis C evidenced by hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis B virus (HBV)-DNA positivity or hepatitis C virus (HCV)-RNA viral load positivity, respectively.
* Negative viral load assays in 2 samples, collected at least 6 months apart, will be required to be considered negative. Both natural clearers and those who have cleared HCV on antiviral therapy are eligible. Participant has an active viral infection based on clinical observation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2035-02-28 (Estimated); Study Completion 2035-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability over time | Up to month 120
  Frequency of adverse events (AEs), serious adverse events (SAEs), and changes from baseline in relevant clinical laboratory tests
GAA enzymatic activity | Baseline and Week 12
  Change from baseline in GAA enzymatic activity in muscle biopsies at week 12
GAA protein expression | Baseline and Week 12
  Change from baseline in GAA protein expression in muscle biopsies at week 12.

SECONDARY OUTCOMES:
Vector Copy Number | Baseline and Week 12
  Change from baseline in vector copy number (VCN) in muscle biopsies at week 12
Thigh Fat Fraction | Baseline and Month 18
  Change from baseline in thigh fat fraction by MRI
6-Minute Walk Test (for ambulatory patients) | Baseline, Week 24 and Week 48
  Change from baseline in the distance walked in the 6 minute walk test (6MWT), which is a standardized assessment of how far an individual can walk on a hard, flat surface in a period of 6 minutes
Percentage Predicted for 6-Minute Walk Test (for ambulatory patients) | Baseline, Week 24 and Week 48
  Change from baseline in percentage predicted for 6MWT, which is a standardized assessment of how far an individual can walk on a hard, flat surface in a period of 6 minutes
Forced Vital Capacity (FVC) | Baseline, Week 24 and Week 48
  Change from baseline in percentage of predicted FVC measured by pulmonary function testing
Maximum Inspiratory Pressure (MIP) | Baseline, Week 24 and Week 48
  Change from baseline in MIP measured by pulmonary function testing
Maximum Expiratory Pressure (MEP) | Baseline, Week 24 and Week 48
  Change from baseline in MEP measured by pulmonary function testing
The Gait, Stairs, Gower Maneuver, Chair (GSGC) | Baseline, Week 24 and Week 48
  The GSGC is a composite test that evaluates both the time to perform different motor activities and qualitatively measures motor function.
Rasch-built Pompe-specific Activity (R-PAct) scale | Baseline and Week 48
  Change from baseline in the R-PAct scale, which was developed to measure Pompe patients' ability carry out daily life activities and social participation
EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) Questionnaire | Baseline and Week 48
  Change from baseline in health profiles and overall health status as assessed by the EQ-5D-5L
Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline and Week 48
  Change from baseline in scores of PROMIS short forms for fatigue, physical function, social participation and sleep disturbance

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- United States (3):
  - University of California Irvine, Department of Neurology, Orange, California
  - Stanford University, Palo Alto, California
  - University of Utah, Division of Medical Genetics, Salt Lake City, Utah
- Newcastle Upon Tyne Hospitals Foundation Trust Clinical Research Facility, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.